CLINICAL TRIAL: NCT00354575
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel Study on the Efficacy and Safety of Traditional Chinese Medicines for Chronic Constipation Residents in Long-Term Care Units
Brief Title: Effect of Chinese Herb on Chronic Constipation for Residents in Long-Term Care Units
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chien-Hsun Huang, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 941216
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-07

CONDITIONS: Chronic Constipation
Keywords: Constipation;; Chinese herb;; Long-term care;; Integrative Chinese Medicine and Western Medicine;
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Chinese Herb (CCH1)
  Interventions: Drug: Chinese Herb: CCH1
- B (Placebo Comparator): Starch powder as placebo
  Interventions: Drug: Chinese Herb: CCH1

INTERVENTIONS:
Drug: Chinese Herb: CCH1 — 1.5/3.0/4.5gm powder per day for mild/moderate/severe constipation

SUMMARY:
The purpose of our study is to improve the problem of constipation and increase the quality of long-term care by the regimen of Chinese herb prescribed by professional doctors of Chinese medicine.

DETAILED DESCRIPTION:
Although many people regard regular defecation as important factor to maintain healthy, constipation is still a common problem in general population. According to some surveys, constipation affects approximately 50% to 73% of nursing home residents. Because the symptoms cause serious impairment of life quality, laxatives are commonly prescribed for people and over-prescribing of laxatives is also common. Despite the large sums spent on laxatives, there have been few advances in laxative treatment in the last 50 years and there have been minimal research addressing the problem. Therefore constipation was labeled as "the neglected symptoms".

There is unsatisfactory effect by currently pharmacologic therapies and preventive strategies for constipation. Contrarily, they had abundant clinical experiences and medical records for constipation in traditional Chinese medicine. So we follow the worldly trend to do the research of integrative Chinese medicine and western medicine since WHO launched the first global strategy on traditional and complementary/alternative medicine (TM/CAM) to assist countries to create a stronger evidence base on the safety, efficacy and quality of the TM/CAM products and practices. The aim of our study is to improve the problem of constipation and increase the quality of long-term care by the regimen of Chinese herb prescribed by professional doctors of Chinese medicine.

The study will be performed under randomized, double-blind, placebo controlled, parallel design. The object of this study is the residents in nursing homes. After intake of Chinese herb, improving constipation and life quality, decreasing the frequency of enema or digital maneuver, minimizing the dosage of laxatives and saving the medical expenditure will be expected.

ELIGIBILITY:
Inclusion Criteria:

* men and non-pregnant women who are at least 20 years of age;
* patients who have been adequately informed of the nature and risks of the study and who have given written informed consent prior to receiving study medication
* residents in long-term care units who meet one of the following criteria in past one month: 1. MgO >= 1 tab tid 2.Dulcolax >=1 tab qd 3.concurrent use of at least two categories of laxatives 4.at least once a week of enema 5.less than three times a week of bowel movement

Exclusion Criteria:

* known renal or hepatic insufficiency;
* known colorectal cancer, anal abscess, anal fistula, anal fissure, rectocele, inflammatory bowel diseases, or gastrointestinal obstruction;
* unknown cause of gastrointestinal bleeding or acute infection
* history of alcohol or drug abuser
* history of psychiatric disorders
* women who are pregnant, as determined by a urine pregnancy test
* use of an investigational drug (within 30days prior to enrollment)
* known allergies to the component of study medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
frequency of spontaneous bowel movement | every week
frequency of enema/digital maneuver every week | every week
amount of rescue laxative use | every week

SECONDARY OUTCOMES:
stool consistency | every week
stool amount | every week
efficacy of treatment evaluated by care-giver | 2 month
evaluation of safety | every week

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsun Huang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Yun-Lin Branch, Douliu, Taiwan

REFERENCES:
- [Background] Lembo A, Camilleri M. Chronic constipation. N Engl J Med. 2003 Oct 2;349(14):1360-8. doi: 10.1056/NEJMra020995. No abstract available. PMID 14523145